CLINICAL TRIAL: NCT00548327
Title: Randomized, Double-Blinded, Placebo Controlled Study of the Effects of Atomoxetine on Cognitive Function in Patients With Schizophrenia and Normal Controls Based on COMT Genotype
Brief Title: The Effects of Atomoxetine on Cognition and Brain Function Based on Catechol-O-methyltransferase(COMT) Genotype
Acronym: Atomoxetine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The scientific director decided to terminate: low priority study with slow accrual
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 080002; Atomoxetine Protocol; Atomoxetine (Other Grant/Funding Number: National Institute of Mental Health); 08-M-0002
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Results first posted 2013-06-14 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-04

CONDITIONS: Schizophrenia; Memory Disorders; Cognition Disorders
Keywords: Genes; Dorsolateral Prefrontal Cortex; Dopamine; Functional Magnetic Resonance Imaging; Neuropsychological Testing; Schizophrenia; Atomoxetine; Cognitive Study; Pharmacogenetics; Normal Volunteers; Catechol-O-Methyltransferase; Healthy Volunteer
MeSH Terms: conditions — Schizophrenia; Memory Disorders; Cognition Disorders | interventions — Atomoxetine Hydrochloride; Neuropsychological Tests

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Active Comparator): Atomoxetine 80 mg final dose. Arm lasts 14 days.
  Schedule 25 mg Day 1 (or Day 22), 40 mg Day 2-3 (or Days 23-24), 60 mg Days 4-5 (or Days 25-26), 80 mg Days 6-14 (or Days 27-35).
  After 14 days, subjects undergo functional magnetic resonance imaging (MRI) and neuropsychological testing in addition to psychopathology ratings
  Interventions: Drug: Atomoxetine; Procedure: Functional magnetic resonance imaging; Procedure: Neuropsychological Testing
- Placebo (Placebo Comparator): Placebo administered for 14 days. Schedule Atomoxetine 25 mg Placebo Day 1 (or Day 22), Atomoxetine 40 mg Placebo Day 2-3 (or Days 23-24), Atomoxetine 60 mg Placebo Days 4-5 (or Days 25-26), Atomoxetine 80 mg Placebo Days 6-14 (or Days 27-35).
  After 14 days, subjects undergo functional magnetic resonance imaging and neuropsychological testing in addition to psychopathology ratings
  Interventions: Procedure: Functional magnetic resonance imaging; Procedure: Neuropsychological Testing; Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Comparison between Atomoxetine and Placebo
  Other Names: Strattera
  Arms: Atomoxetine
Procedure: Functional magnetic resonance imaging — Comparison between Atomoxetine and Placebo arms
Procedure: Neuropsychological Testing — Comparison between Atomoxetine and Placebo arms
  Other Names: Neuropsychiatric testing
Drug: Placebo — 25 mg, 40 mg, 60 mg and 80 mg Atomoxetine Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate whether Atomoxetine improves cognition in healthy volunteers as well as patients with schizophrenia. Atomoxetine is a drug that has been Food and Drug Administration (FDA) approved for Attention Deficit Disorder and allegedly increase the amount of the neurotransmitter dopamine in the frontal cortex of the brain.

DETAILED DESCRIPTION:
Psychopharmacological modulation of the catecholaminergic system can enhance some aspects of cognitive function. For example, catechol-O-methyltransferase (COMT) inhibitors such as tolcapone can improve working memory/executive function. Similarly, modafinil, a catecholaminergic agonist with norepinephrine (NA) reuptake blocking properties, was also shown to improve delay-dependent working memory in mice. Differences in the response between individuals might be related to a number of factors, including variations in the genes. The recent finding that a polymorphism in the COMT gene, which produces a change in enzyme activity, accounts for 4% of the variance in performance of working memory tasks in humans suggest that COMT genotype may predict response to COMT inhibitors or to other dopaminergic agonists that increase catecholaminergic function in the frontal cortex. In the present investigation our goal is to examine, in normal controls and patients with schizophrenia, the effect of atomoxetine, a selective noradrenaline reuptake inhibitor that increases extracellular levels of dopamine in the frontal cortex, on cognitive function. We predict that both normal controls and patients with schizophrenia with the val/val genotype, which present higher COMT activity and, thus, lower extracellular dopamine concentrations in the frontal cortex, will have a significant improvement in working memory. Furthermore, in conjunction with other National Institute of Mental Health imaging protocols, we would like to examine the neurophysiological correlates related to working memory. We predict improved measures in prefrontal efficiency in subjects and patients specifically with the val/val genotype. The present protocol will provide new insights on the importance of this genetic polymorphism in the regulation of aminergic-controlled cognitive function in normal individuals. Furthermore, this protocol will test whether atomoxetine offers a new treatment, based on genotype, for cognitive impairment in schizophrenia. An Investigational New Drug (IND) waiver will be requested for the present study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Prior participation under NIH protocol # 95-M-0150, or new normal volunteers or schizophrenic patients that meet criteria for NIH protocol # 95-M-0150.
* No active Axis I or Axis II diagnosis in normal volunteers.
* Age range: 18-45 years.
* Normal EKG and blood pressure readings.

EXCLUSION CRITERIA:

* Normal volunteers with an active Axis I or Axis II disorder or patients with an Axis I diagnosis other than schizophrenia or schizoaffective disorder obtained either from prior Structured Clinical Interview for the Diagnostic and Statistical Manual Disorders (SCID) interview in Protocol 95-M-0150 or through a screening interview will be excluded.
* Subjects with a history of cardiovascular disease, liver disease and other serious medical illnesses, and untreated or uncontrolled hypertension will be excluded because of the potential for drug-drug interaction or because of the potential deleterious effect of the drug on the medical condition. An electrocardiogram, blood pressure, pulse rate, toxicological screen, cell blood count and metabolic panel including Liver Function Tests (LFTs) will be checked on all subjects prior to participation in the study. Any subject with an electrocardiogram deemed abnormal by a cardiologist or with sustained systolic blood pressure of 150 mmHg or above, diastolic blood pressure of 100 mmHg or above will be excluded from the study.
* Schizophrenic patients taking a COMT inhibitor, any illicit drugs of abuse, or Monoamine Oxidase (MAO) inhibitors will be excluded. Patients taking paroxetine, fluoxetine, bupropion, tricyclic antidepressants, albuterol, modafinil, stimulants or pressor agents will be excluded from the study. No medication will be stopped in order to participate in the study.
* Normal control subjects taking any medication other than occasional nonsteroidal anti-inflammatory drugs (NSAID) or with recent history of illicit drug or alcohol abuse will be excluded. Normal controls on contraceptive medication will be excluded from the study.
* Pregnant women: Women of childbearing potential will undergo a urine pregnancy test the day the study initiates and they will be screened by history for the possibility of pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2007-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Apud, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Beracochea D, Cagnard B, Celerier A, le Merrer J, Peres M, Pierard C. First evidence of a delay-dependent working memory-enhancing effect of modafinil in mice. Neuroreport. 2001 Feb 12;12(2):375-8. doi: 10.1097/00001756-200102120-00038. PMID 11209953
- [Background] Egan MF, Goldberg TE, Kolachana BS, Callicott JH, Mazzanti CM, Straub RE, Goldman D, Weinberger DR. Effect of COMT Val108/158 Met genotype on frontal lobe function and risk for schizophrenia. Proc Natl Acad Sci U S A. 2001 Jun 5;98(12):6917-22. doi: 10.1073/pnas.111134598. Epub 2001 May 29. PMID 11381111
- [Background] de Saint Hilaire Z, Orosco M, Rouch C, Blanc G, Nicolaidis S. Variations in extracellular monoamines in the prefrontal cortex and medial hypothalamus after modafinil administration: a microdialysis study in rats. Neuroreport. 2001 Nov 16;12(16):3533-7. doi: 10.1097/00001756-200111160-00032. PMID 11733706
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-M-0002.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Normal volunteers or patients with schizophrenia will be initially recruited from among individuals who have volunteered for previous genetic studies and for whom genetic data is already available. Power calculations set target accrual at 30 participants per genotype for 3 COMT genotypes per cohort (i.e., 90 patients and 90 healthy volunteers).
Pre-assignment Details: Subjects need to satisfy the inclusion/exclusion criteria for the genetic studies protocol before participating. Normal volunteers will be enrolled as outpatients and patients as inpatients. Females do both arms during the same phase of the menstrual cycle. Patients with Schizophrenia are stabilized for at least 6 weeks before the protocol.
Groups:
- Healthy Participants: This is a double-blind, placebo-control, cross-over study of Atomoxetine in healthy volunteers. It includes 3 genotypes, the VAL/VAL, VAL/MET and MET/MET. Subjects are 2 weeks on placebo, 2 weeks on active compound and one week wash-out period between arms.
  Amoxetine schedule: 25 mg Day 1 (or Day 22), 40 mg Day 2-3 (or Days 23-24), 60 mg Days 4-5 (or Days 25-26), 80 mg Days 6-14 (or Days 27-35).
  Placebo schedule: Atomoxetine 25 mg Placebo Day 1 (or Day 22), Atomoxetine 40 mg Placebo Day 2-3 (or Days 23-24), Atomoxetine 60 mg Placebo Days 4-5 (or Days 25-26), Atomoxetine 80 mg Placebo Days 6-14 (or Days 27-35).
- Patients With Schizophrenia: This is a double-blind, placebo-control, cross-over study of Atomoxetine in patients with schizophrenia. It includes 3 genotypes, the VAL/VAL, VAL/MET and MET/MET. Subjects are 2 weeks on placebo, 2 weeks on active compound and one week wash-out period between arms.
  Amoxetine schedule: 25 mg Day 1 (or Day 22), 40 mg Day 2-3 (or Days 23-24), 60 mg Days 4-5 (or Days 25-26), 80 mg Days 6-14 (or Days 27-35).
  Placebo schedule: Atomoxetine 25 mg Placebo Day 1 (or Day 22), Atomoxetine 40 mg Placebo Day 2-3 (or Days 23-24), Atomoxetine 60 mg Placebo Days 4-5 (or Days 25-26), Atomoxetine 80 mg Placebo Days 6-14 (or Days 27-35).
Period: Overall Study
Arm/Group | Healthy Participants | Patients With Schizophrenia
Started | 6 | 5
Completed | 6 | 4 (Patient randomized to receive placebo first. While on placebo, Adverse Event lead to discontinuation)
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Patients With Schizophrenia | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 45 years | 6 | 5 | 11
  >=45 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Changes in Functional Magnetic Resonance Imaging (fMRI) Blood-oxygen-level-dependent (Bold) Activity
Description: Main outcome measures were BOLD fMRI response (activation) while performing a prefrontal cortex-dependent task such as N-Back Working Memory with increasing levels of task difficulty. It was expected to have a greater level of activation in BOLD fMRI in schizophrenic patients with respect to normal volunteers, and a greater activation in individuals (either normal volunteers or patients) who share the val/val genotype with respect to the met/met genotype.
  Based on prior fMRI studies and on power analysis of neuropsychological variables, at least 28 and 26 subjects are respectively needed to achieve significant power in functional neuroimaging and neuropsychological studies.These sizes provide an 80% power to observe significant differences between drug conditions at the 0.05 level.
Time Frame: 2 hours after the first or the second dose of Atomoxetine or placebo on 14th day
Population: Data were not collected for analysis because the study was terminated before target accrual
Arm/Group | Healthy Participants | Patients With Schizophrenia
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in The Positive and Negative Syndrome Scale (PANSS)
Description: The Positive and Negative Syndrome Scale (PANSS) is a 7-point rating scale with (1) indicating the absence of a symptom or behavior and (7) indicating the most severe symptom. The PANSS includes three scales(Positive and Negative Syndromes and General Psychopathology)and five clusters (Anergia, Thought Disturbance, Activation, Paranoid/Belligerence and Depression.
Time Frame: At 14th and 35th days
Population: Data were not collected for analysis because the study was terminated before target accrual
Arm/Group | Healthy Participants | Patients With Schizophrenia
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Changes in Cognitive Function Measured by Neuropsychological Testing
Description: Neuropsychological testing consists of a battery of 10-12 individual tests to measure cognitive function. We expect both a drug effect and a genotype effect on neuropsychological tasks that measure dorsolateral prefrontal cortex (DLPFC) executive function, mostly in individuals who share the val/val genotype with respect to the met/met genotype.
Time Frame: 2 hours after the first or the second dose of Atomoxetine or placebo on 14th day
Population: Data were not collected for analysis because the study was terminated before target accrual
Arm/Group | Healthy Participants | Patients With Schizophrenia
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in The Profile of Mood States
Description: The Profile of Mood States is an instrument that provides a rapid method of assessing transient, fluctuating mood states. The POMS consists of 65 adjectives rated by subjects on a 5-point scale and six factors that derive from this scale are: 1)tension-anxiety, 2)depression-dejection, 3)anger-hostility, 4)fatigue-inertia, 5)vigor-activity and 6)Confusion-bewilderment.
Time Frame: At 14th and 35th days
Population: Data were not collected for analysis because the study was terminated before target accrual
Groups:
- Healthy Participants: Atomoxetine 40 mg twice daily (bid), placebo, Val/Val, Val/Met, Met/Met.
Arm/Group | Healthy Participants | Patients With Schizophrenia
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in The Hamilton Anxiety Rating Scale
Description: The Hamilton Anxiety Rating Scale is a psychological questionnaire to rate the severity of anxiety.It contains 14 symptom-oriented questions.Each of these symptoms is given a severity rating, from not present(scored as 0)to very severe(scored as 4)
Time Frame: At 14th and 35th days
Population: Data were not collected for analysis because the study was terminated before target accrual
Arm/Group | Healthy Participants | Patients With Schizophrenia
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Blood Plasma Concentration of Atomoxetine
Description: Blood for drug plasma levels is obtained before and 3 hours after dosing on the 14th day receiving Atomoxetine.
Time Frame: before and 3 hours after dosing on the 14th day receiving Atomoxetine
Population: Data were not collected for analysis because the study was terminated before target accrual
Arm/Group | Healthy Participants | Patients With Schizophrenia
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Two years, from 2008 to 2011.
Description: Adverse events are collected during the arm or at the end of each arm.
Arm/Group | Atomoxetine-Patient | Placebo-Patient | Atomoxetine-Healthy Volunteer | Placebo-Healthy Volunteer
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/5 | 2/5 | 4/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine-Patient (N=5) | Placebo-Patient (N=5) | Atomoxetine-Healthy Volunteer (N=6) | Placebo-Healthy Volunteer (N=6)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine-Patient (N=5) | Placebo-Patient (N=5) | Atomoxetine-Healthy Volunteer (N=6) | Placebo-Healthy Volunteer (N=6)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Mild. Present in both arms of the protocol in one patient
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Mild
Difficulty sleeping (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) — Mild. Present in both arms of the protocol in one healthy volunteer and one patient
Loss of Appetite (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) — Mild in two patients,one of them on placebo and moderate in one HV
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 1 (1) — Two patients had the side effect during both arms of the protocol
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) — One subject had the side effect in both arms of the protocol.
Fatigue (Psychiatric disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1) — Fatigue was present in 2 patients and 1 HV in both arms of the protocol.
Sexual dysfuntion (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Side effect was present in both arms of the protocol in one patient
Urinary difficulties (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mild
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Side effect present in both arms of the protocol in one patient
Restlessness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Side effect present in both arms of the protocol in one patient
Heartburn (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Side effect present in one patient in both arms of the protocol
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
unusual thoughts (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No